CLINICAL TRIAL: NCT03304873
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of the Efficacy of Retapamulin as a Topical Decolonizing Agent for Mupirocin Resistant Methicillin Resistant Staphylococcus Aureus (MRSA)
Brief Title: Retapamulin as a Decolonizing Agent for MRSA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-00907
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: MRSA
Keywords: rectal MRSA; mupirocin-resistant nasal MRSA
MeSH Terms: interventions — retapamulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Retapamulin (Experimental): Thin layer of ointment applied twice a day for five days. Study drug will be applied to the nares and peri-rectal area twice a day for 5 consecutive days.
  Interventions: Drug: Retapamulin
- Placebo (Placebo Comparator): The placebo used will be a triple purified pharmaceutical grade white petrolatum
  Interventions: Drug: Placebo Ointment

INTERVENTIONS:
Drug: Retapamulin — Retapamulin is a topical antibiotic ointment. The ingredients include retapamulin and white petrolatum as the vehicle. The composition is 10mg retapamulin per 1g of ointment (1%).
  Arms: Retapamulin
Drug: Placebo Ointment — The placebo that will be used is triple-purified pharmaceutical-grade petrolatum.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy of retapamulin to reduce carriage of MRSA via a randomized, double-blind, placebo-controlled clinical study testing retapamulin among patients with confirmed mupirocin-resistant nasal and/or rectal MRSA colonization. The sample size will include 27 subjects in each of the two arms of the study (retapamulin versus placebo) for a total of 54 subjects. Participants who are found to be nasal and/or rectal colonized with MRSA will be randomized to receive either retapamulin or placebo applied nasally and rectally for a total of 5 days. Nasal and rectal swabs will be collected at pre-defined time points during study duration (screening swab, swab one week after completion of topical therapy, swab 4 weeks after completion of topical therapy) to assess MRSA colonization status. The colonization rates of both groups will be assessed via Fisher's Exact Test.

ELIGIBILITY:
Inclusion Criteria:

1. Admission to the general pediatric floor and pediatric intensive care units at NYU Langone Medical Center or visit to study team members at ODA clinic (Park Ave locations) in Williamsburg Brooklyn.
2. Ages 9 months to 17 years
3. Residing in the zip codes which reflect Orthodox Jewish neighborhoods where there is a current outbreak of this strain of MRSA.
4. Nasal and/or rectal culture positive for mupirocin-resistant methicillin-resistant Staphylococcus aureus (MRSA)

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pregnant or lactating
2. Unable to appropriately consent
3. Open sores in either of the study sites (nares or rectum)
4. Recent surgical procedure to either study site (nares or rectum)
5. Concurrent use of Rifampin or Trimethoprim/Sulfamethoxazole
6. Current active MRSA infection
7. Immunocompromised
8. Presence of endotracheal tube, tracheostomy tube or other foreign body in upper airway

Ages: 9 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Lighter, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Retapamulin | Placebo
Started | 23 | 24
Completed | 22 | 16
Not Completed | 1 | 8
Not completed — Lost to Follow-up | 1 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retapamulin | Placebo | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Median (Full Range); unit: years] | 3.9 [0.75 to 12] | 3.5 [0.75 to 14] | 3.5 [0.75 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 28
  Male | 5 | 14 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With MRSA Carriage at 1 Week Post Decolonization With Retapamulin or Placebo
Description: Study visit for nasal/peri-rectal swabs
Time Frame: 1 Week
Measure: Count of Participants; unit: Participants
Arm/Group | Retapamulin | Placebo
Number analyzed (Participants) | 23 | 22
Participants | 2 | 13
Statistical Analysis 1: Comparison: Retapamulin vs Placebo; Test type: Superiority; p = 0.0004, t-test, 1 sided

2. Primary Outcome: Number of Partcipants With MRSA Carriage at 4 Weeks Post Decolonization With Retapamulin or Placebo
Description: Study visit for nasal/peri-rectal swabs
Time Frame: 4 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Retapamulin | Placebo
Number analyzed (Participants) | 22 | 16
Participants | 12 | 9
Statistical Analysis 1: Comparison: Retapamulin vs Placebo; Test type: Superiority; p = 0.99, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: While on study protocol, which includes while using randomized medication and throughout follow-up (about 6 weeks).
Description: Known risks or adverse reactions from this drug use are minimal and include local application site irritation (pruritus, erythema, stinging). In clinical studies, this was found to occur in < 2% of patients. This information is listed in the package insert for retapamulin. It is expected not to pose greater than minimal risk to participants. Side effects of Retapamulin are not commonly expected and are reported to subside with the discontinuation of the drug without expected long term risks.
Arm/Group | Retapamulin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 14/23 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retapamulin (N=23) | Placebo (N=24)
Local application site irritation (General disorders) | 14 (14) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT03304873/Prot_SAP_000.pdf